CLINICAL TRIAL: NCT01115738
Title: TRansferring From ClopIdogrel Loading Dose to Prasugrel Loading Dose in Acute Coronary Syndrome PatiEnTs: TRIPLET
Brief Title: Clopidogrel to Prasugrel in Acute Coronary Syndrome (ACS) Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13533; H7T-CR-TAEH (Other: Eli Lilly and Company); CTRI/2010/091/000348 (Registry Identifier: India)
Record Dates: First submitted 2010-04-23; First posted 2010-05-04 (Estimated); Results first posted 2012-10-26 (Estimated); Last update posted 2012-11-20 (Estimated); Status verified 2012-11

CONDITIONS: Acute Coronary Syndrome
Keywords: Plavix, Effient
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Prasugrel Hydrochloride; Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo and 60 milligram (mg) Prasugrel (Placebo Comparator): Placebo loading dose administered once orally before percutaneous coronary intervention (PCI) and 60-mg prasugrel loading dose administered once orally during PCI, followed by 10-mg prasugrel maintenance dose administered orally 24 hours after loading dose, then every 24 hours for 72 hours.
  Interventions: Drug: Prasugrel; Drug: Placebo
- 600 mg Clopidogrel and 60 mg Prasugrel (Experimental): 600-mg clopidogrel loading dose administered once orally before PCI and 60-mg prasugrel loading dose administered once orally during PCI, followed by 10-mg prasugrel maintenance dose administered orally 24 hours after loading dose, then every 24 hours for 72 hours.
  Interventions: Drug: Prasugrel; Drug: Clopidogrel
- 600 mg Clopidogrel and 30 mg Prasugrel (Experimental): 600-mg clopidogrel loading dose administered once orally before PCI and 30-mg prasugrel loading dose administered once orally during PCI, followed by 10-mg prasugrel maintenance dose administered orally 24 hours after loading dose, then every 24 hours for 72 hours.
  Interventions: Drug: Prasugrel; Drug: Clopidogrel

INTERVENTIONS:
Drug: Prasugrel — Loading dose administered once orally and maintenance dose administered orally 24 hours after loading dose, then every 24 hours for 72 hours.
  Other Names: LY640315
Drug: Clopidogrel — Loading dose administered once orally.
  Arms: 600 mg Clopidogrel and 30 mg Prasugrel; 600 mg Clopidogrel and 60 mg Prasugrel
Drug: Placebo — Loading dose administered once orally
  Arms: Placebo and 60 milligram (mg) Prasugrel

SUMMARY:
This study will evaluate the use of a prasugrel 60 mg loading dose (LD) administered during percutaneous coronary intervention (PCI) with and without a prior LD of clopidogrel on platelet inhibition in patients presenting with acute coronary syndrome (ACS). Platelet inhibition following a prasugrel LD in clopidogrel pretreated patients' will be determined in a time-dependent manner for two different prasugrel loading doses (30 mg and 60 mg). Understanding the effects of this combination on platelet inhibition will provide guidance to physicians on the use of prasugrel in patients who have already been pretreated with clopidogrel.

ELIGIBILITY:
Inclusion Criteria:

* Participants hospitalized with acute coronary syndrome (ACS) [unstable angina (UA), non-ST elevation myocardial infarction (NSTEMI), or ST elevation myocardial infarction (STEMI)] as determined by the investigator, and who are anticipated to undergo percutaneous coronary intervention (PCI) as a treatment for the ACS event within 24 hours of the clopidogrel/placebo loading dose
* Participants provide signed informed consent form (ICF)
* Participants weigh at least 60 kilograms (kg) at the time of screening
* Women of child-bearing potential (that is, women who are not surgically or chemically sterilized and who are between menarche and 1-year postmenopause), test negative for pregnancy at the time of enrollment based on a urine or serum pregnancy test

Exclusion Criteria:

* Have cardiogenic shock at the time of randomization (systolic blood pressure greater than 90 millimeters of mercury (mm Hg) associated with clinical evidence of end-organ hypoperfusion, or participants requiring vasopressors to maintain systolic blood pressure over 90 mm Hg and associated with clinical evidence of end-organ hypoperfusion
* Have refractory ventricular arrhythmias
* Have New York Heart Association (NYHA) Class IV congestive heart failure
* Have systolic blood pressure greater than 180 mm Hg, or diastolic blood pressure greater than 100 mm Hg on more than 1 assessment at any time from participant presentation of ACS treatment to enrollment
* Have received fibrin-specific fibrinolytic therapy less than 24 hours prior to randomization
* Have received nonfibrin-specific fibrinolytic therapy less than 48 hours prior to randomization
* Have active internal bleeding or history of bleeding diathesis
* Have clinical findings, in the judgment of the investigator, associated with an increased risk of bleeding
* Prior history of ischemic or hemorrhagic stroke
* Intracranial neoplasm, arteriovenous malformation, or aneurysm
* Prior history of transient ischemic attack (TIA)
* Have an International Normalized Ratio (INR) known to be greater than 1.5 at the time of evaluation
* Have a platelet count of less than 100,000 per cubic millimeter (mm^3) at the time of evaluation
* Have anemia [hemoglobin (Hgb) less than 10 grams per deciliter (g/dL)] at the time of evaluation
* Have received 1 or more doses of a thienopyridine (ticlopidine, clopidogrel, or prasugrel) or other adenosine diphosphate (ADP) receptor inhibitor within 10 days prior to screening
* Have been administered glycoprotein IIb/IIIa (GPIIb/IIIa) inhibitor within the past 7 days or planned use of a GPIIb/IIIa inhibitor during PCI
* Are receiving or will receive oral anticoagulation or other antiplatelet therapy, other than aspirin (ASA), which cannot be safely discontinued for the duration of the study.
* Are receiving daily treatment with nonsteroidal anti-inflammatory drugs (NSAIDs) or cyclooxygenase-2 (COX2) inhibitors that cannot be discontinued during the study
* Are currently enrolled in, or discontinued within the last 30 days from, a clinical trial involving an investigational drug or device or off-label use of a drug or device, or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Have previously completed or withdrawn from this study or any other study investigating prasugrel
* Are women who are known to be pregnant, who have given birth within the past 90 days, or who are breastfeeding
* Have a concomitant medical illness (for example, terminal malignancy) that in the opinion of the investigator, is associated with reduced survival over the expected treatment period
* Have known severe hepatic dysfunction (that is, with cirrhosis or portal hypertension)
* Have a history of intolerance or allergy to aspirin or approved thienopyridines (ticlopidine, clopidogrel or prasugrel)
* May be unable to cooperate with protocol requirements and follow-up procedures

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2010-05; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- India (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bangalore
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyderabaad
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Delhi

REFERENCES:
- [Derived] Diodati JG, Saucedo JF, Cardillo TE, Jakubowski JA, Henneges C, Effron MB, Lipkin FR, Walker JR, Duvvuru S, Sundseth SS, Fisher HN, Angiolillo DJ. Transferring from clopidogrel loading dose to prasugrel loading dose in acute coronary syndrome patients. High on-treatment platelet reactivity analysis of the TRIPLET trial. Thromb Haemost. 2014 Aug;112(2):311-22. doi: 10.1160/TH13-09-0747. Epub 2014 Apr 10. PMID 24718367
- [Derived] Diodati JG, Saucedo JF, French JK, Fung AY, Cardillo TE, Henneges C, Effron MB, Fisher HN, Angiolillo DJ. Effect on platelet reactivity from a prasugrel loading dose after a clopidogrel loading dose compared with a prasugrel loading dose alone: Transferring From Clopidogrel Loading Dose to Prasugrel Loading Dose in Acute Coronary Syndrome Patients (TRIPLET): a randomized controlled trial. Circ Cardiovasc Interv. 2013 Oct 1;6(5):567-74. doi: 10.1161/CIRCINTERVENTIONS.112.000063. Epub 2013 Sep 24. PMID 24065443

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo and 60-mg Prasugrel: Placebo loading dose (LD) administered once orally before percutaneous coronary intervention (PCI) and 60-milligram (mg) prasugrel LD administered once orally during PCI, followed by 10-mg prasugrel maintenance dose administered orally 24 hours after LD, then every 24 hours for 72 hours.
- 600-mg Clopidogrel and 60-mg Prasugrel: 600-mg clopidogrel LD administered once orally before PCI and 60-mg prasugrel LD administered once orally during PCI, followed by 10-mg prasugrel maintenance dose administered orally 24 hours after LD, then every 24 hours for 72 hours.
- 600-mg Clopidogrel and 30-mg Prasugrel: 600-mg clopidogrel LD administered once orally before PCI and 30-mg prasugrel LD administered once orally during PCI, followed by 10-mg prasugrel maintenance dose administered orally 24 hours after LD, then every 24 hours for 72 hours.
Period: Overall Study
Arm/Group | Placebo and 60-mg Prasugrel | 600-mg Clopidogrel and 60-mg Prasugrel | 600-mg Clopidogrel and 30-mg Prasugrel
Started | 110 | 83 | 89
Received Any Treatment | 109 | 79 | 88
Pharmacodynamic (PD) Population | 52 (Received prasugrel LD and had at least one evaluable PD measurement after prasugrel LD.) | 47 (Received prasugrel LD and had at least one evaluable PD measurement after prasugrel LD.) | 50 (Received prasugrel LD and had at least one evaluable PD measurement after prasugrel LD.)
Completed | 85 | 62 | 62
Not Completed | 25 | 21 | 27
Not completed — Death | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Physician Decision | 18 | 15 | 17
Not completed — Withdrawal by Subject | 6 | 6 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo and 60-mg Prasugrel | 600-mg Clopidogrel and 60-mg Prasugrel | 600-mg Clopidogrel and 30-mg Prasugrel | Total
Number analyzed (Participants) | 52 | 47 | 50 | 149
Age Continuous [Mean (Standard Deviation); unit: years] | 58.1 (9.47) | 57.5 (9.12) | 58.7 (8.07) | 58.1 (8.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 8 | 9 | 30
  Male | 39 | 39 | 41 | 119
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 14 | 13 | 40
  Not Hispanic or Latino | 30 | 28 | 30 | 88
  Unknown or Not Reported | 9 | 5 | 7 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 13 | 12 | 9 | 34
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 0 | 3
  Black or African American | 1 | 2 | 3 | 6
  White | 37 | 31 | 38 | 106
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  India | 10 | 11 | 9 | 30
  Argentina | 2 | 4 | 4 | 10
  Brazil | 6 | 5 | 6 | 17
  Australia | 1 | 3 | 2 | 6
  Canada | 11 | 8 | 10 | 29
  Mexico | 8 | 6 | 5 | 19
  Turkey | 7 | 2 | 7 | 16
  United States | 7 | 8 | 7 | 22
Qualifying Acute Coronary Syndrome (ACS) Event [Number; unit: participants]
  Unstable Angina | 21 | 16 | 22 | 59
  Non-ST-elevation Myocardial Infarction | 20 | 18 | 21 | 59
  ST-elevation Myocardial Infarction | 11 | 13 | 7 | 31

OUTCOME MEASURES:

1. Primary Outcome: Adenosine Diphosphate (ADP)-Induced P2Y12 Receptor-Mediated Platelet Aggregation 6 Hours After Prasugrel Loading Dose (LD)
Description: ADP-induced P2Y12 receptor mediated platelet aggregation serves as a biomarker of platelet function. It is measured in P2Y12 Reaction Units (PRU) with lower PRU reflecting stronger inhibition of P2Y12 and reduced platelet aggregation. Least Squares (LS) Mean values were controlled for treatment, visit, treatment and visit interaction, and country.
Time Frame: 6 hours after prasugrel loading dose
Population: All randomized participants who received the prasugrel LD and had at least one evaluable PRU measurement after LD.
Measure: Least Squares Mean (Standard Error); unit: PRU
Arm/Group | Placebo and 60-mg Prasugrel | 600-mg Clopidogrel and 60-mg Prasugrel | 600-mg Clopidogrel and 30-mg Prasugrel
Number analyzed (Participants) | 52 | 47 | 50
PRU | 57.86 (11.86) | 35.61 (12.36) | 53.92 (11.74)
Statistical Analysis 1: Comparison: Placebo and 60-mg Prasugrel vs 600-mg Clopidogrel and 60-mg Prasugrel; Test type: Superiority or Other; p = 0.188, Mixed Model Repeated Measures Analysis — P-values were not adjusted for multiplicity. P-values <0.05 were considered statistically significant; Fixed effects were Treatment, Visit, Country, Treatment-by-Visit. Participants and Error were Random Effects. Covariance structure was Unstructured; Mean Difference (Final Values) = 22.24, 95% CI 2-sided [-10.98 to 55.47]
Statistical Analysis 2: Comparison: Placebo and 60-mg Prasugrel vs 600-mg Clopidogrel and 30-mg Prasugrel; Test type: Superiority or Other; p = 0.809, Mixed Model Repeated Measures Analysis — P-values were not adjusted for multiplicity. P-values <0.05 were considered statistically significant; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 3.93, 95% CI 2-sided [-28.20 to 36.07]

2. Secondary Outcome: Adenosine Diphosphate (ADP)-Induced P2Y12 Receptor-Mediated Platelet Aggregation at Baseline, 2, 24 and 72 Hours After Prasugrel Loading Dose (LD)
Description: as for outcome 1
Time Frame: Baseline and 2 hours and 24 hours and 72 hours after prasugrel loading dose
Population: All randomized participants who received prasugrel LD and had at least one evaluable PRU measurement after prasugrel LD.
Measure: Least Squares Mean (Standard Error); unit: PRU
Arm/Group | Placebo and 60-mg Prasugrel | 600-mg Clopidogrel and 60-mg Prasugrel | 600-mg Clopidogrel and 30-mg Prasugrel
Number analyzed (Participants) | 52 | 47 | 50
PRU
  Baseline | 265.51 (13.01) | 248.58 (13.99) | 229.62 (13.38)
  2 Hours after Prasugrel LD | 122.55 (17.28) | 113.10 (18.07) | 117.10 (17.47)
  24 Hours after Prasugrel LD | 62.73 (10.43) | 34.05 (10.88) | 51.43 (10.72)
  72 Hours after Prasugrel LD | 56.95 (8.40) | 48.08 (9.09) | 60.29 (9.05)
Statistical Analysis 1: Comparison: Placebo and 60-mg Prasugrel vs 600-mg Clopidogrel and 60-mg Prasugrel; Test type: Superiority or Other; p = 0.370, Mixed Model Repeated Measures Analysis — P-value is for Baseline. P-values were not adjusted for multiplicity. P-values <0.05 were considered statistically significant; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 16.93, 95% CI 2-sided [-20.26 to 54.12]
Statistical Analysis 2: Comparison: Placebo and 60-mg Prasugrel vs 600-mg Clopidogrel and 30-mg Prasugrel; Test type: Superiority or Other; p = 0.052, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 35.89, 95% CI 2-sided [-0.29 to 72.06]
Statistical Analysis 3: Comparison: Placebo and 60-mg Prasugrel vs 600-mg Clopidogrel and 60-mg Prasugrel; Test type: Superiority or Other; p = 0.703, Mixed Model Repeated Measures Analysis — P-value is for 2 hours after prasugrel LD. P-values were not adjusted for multiplicity. P-values <0.05 were considered statistically significant; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 9.45, 95% CI 2-sided [-39.55 to 58.45]
Statistical Analysis 4: Comparison: Placebo and 60-mg Prasugrel vs 600-mg Clopidogrel and 30-mg Prasugrel; Test type: Superiority or Other; p = 0.823, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 3]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 5.45, 95% CI 2-sided [-42.53 to 53.44]
Statistical Analysis 5: Comparison: Placebo and 60-mg Prasugrel vs 600-mg Clopidogrel and 60-mg Prasugrel; Test type: Superiority or Other; p = 0.054, Mixed Model Repeated Measures Analysis — P-value is for 24 hours after prasugrel LD. P-values were not adjusted for multiplicity. P-values <0.05 were considered statistically significant; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 28.69, 95% CI 2-sided [-0.47 to 57.84]
Statistical Analysis 6: Comparison: Placebo and 60-mg Prasugrel vs 600-mg Clopidogrel and 30-mg Prasugrel; Test type: Superiority or Other; p = 0.436, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 5]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 11.30, 95% CI 2-sided [-17.29 to 39.90]
Statistical Analysis 7: Comparison: Placebo and 60-mg Prasugrel vs 600-mg Clopidogrel and 60-mg Prasugrel; Test type: Superiority or Other; p = 0.463, Mixed Model Repeated Measures Analysis — P-value is for 72 hours after prasugrel LD. P-values were not adjusted for multiplicity. P-values <0.05 were considered statistically significant; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 8.87, 95% CI 2-sided [-14.96 to 32.71]
Statistical Analysis 8: Comparison: Placebo and 60-mg Prasugrel vs 600-mg Clopidogrel and 30-mg Prasugrel; Test type: Superiority or Other; p = 0.777, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 7]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.34, 95% CI 2-sided [-26.62 to 19.94]

3. Secondary Outcome: Mean Change From Baseline to 72 Hours in Laboratory Measurements - Hematocrit
Time Frame: Baseline, 72 hours
Population: All randomized participants who received prasugrel loading dose (LD) and had a Hematocrit measurement 72 hours after LD.
Measure: Mean (Standard Deviation); unit: proportion of 1.0
Arm/Group | Placebo and 60-mg Prasugrel | 600-mg Clopidogrel and 60-mg Prasugrel | 600-mg Clopidogrel and 30-mg Prasugrel
Number analyzed (Participants) | 43 | 38 | 36
proportion of 1.0 | 0.0 (0.04) | 0.0 (0.03) | 0.0 (0.03)

4. Secondary Outcome: Mean Change From Baseline to 72 Hours in Laboratory Measurements - Hemoglobin
Time Frame: Baseline, 72 hours
Population: All randomized participants who received prasugrel loading dose (LD) and had a Hemoglobin measurement 72 hours after LD.
Measure: Mean (Standard Deviation); unit: gram per deciliter (g/dL)
Arm/Group | Placebo and 60-mg Prasugrel | 600-mg Clopidogrel and 60-mg Prasugrel | 600-mg Clopidogrel and 30-mg Prasugrel
Number analyzed (Participants) | 43 | 38 | 36
gram per deciliter (g/dL) | -0.9 (1.41) | -0.6 (1.03) | -0.6 (1.04)

5. Secondary Outcome: Percentage of Inhibition of Platelet Aggregation
Description: Adenosine Diphosphate (ADP)-induced P2Y12 receptor mediated platelet aggregation serves as a biomarker of platelet function. It is measured in P2Y12 Reaction Units (PRU) with lower PRU reflecting stronger inhibition of P2Y12 and reduced platelet aggregation. The internal BASE standard is an independent measurement and serves as an estimate of the participant's baseline platelet aggregation independent of P2Y12 receptor inhibition. Percent Inhibition of Platelet Aggregation=(1-[PRU/BASE) x 100%, high numbers represent increased platelet inhibition. Least Squares (LS) Mean values were controlled for treatment, visit, treatment and visit interaction, and country.
Time Frame: Baseline and 2 and 6 and 24 and 72 hours after loading dose
Population: All randomized participants who received prasugrel loading dose (LD) and had at least one evaluable PRU measurement after prasugrel LD.
Measure: Least Squares Mean (Standard Error); unit: percentage of inhibition
Arm/Group | Placebo and 60-mg Prasugrel | 600-mg Clopidogrel and 60-mg Prasugrel | 600-mg Clopidogrel and 30-mg Prasugrel
Number analyzed (Participants) | 52 | 47 | 50
percentage of inhibition
  Baseline | 9.71 (3.44) | 13.02 (3.70) | 14.94 (3.54)
  2 Hours after Prasugrel LD | 56.04 (5.88) | 58.75 (6.16) | 54.89 (5.95)
  6 Hours after Prasugrel LD | 79.87 (3.95) | 86.77 (4.13) | 78.55 (3.93)
  24 Hours after Prasugrel LD | 77.57 (3.56) | 87.64 (3.74) | 78.56 (3.68)
  72 Hours after Prasugrel LD | 78.48 (2.95) | 83.51 (3.28) | 78.17 (3.27)
Statistical Analysis 1: Comparison: Placebo and 60-mg Prasugrel vs 600-mg Clopidogrel and 60-mg Prasugrel; Test type: Superiority or Other; p = 0.505, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.31, 95% CI 2-sided [-13.10 to 6.48]
Statistical Analysis 2: Comparison: Placebo and 60-mg Prasugrel vs 600-mg Clopidogrel and 30-mg Prasugrel; Test type: Superiority or Other; p = 0.278, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -5.23, 95% CI 2-sided [-14.74 to 4.27]
Statistical Analysis 3: Comparison: Placebo and 60-mg Prasugrel vs 600-mg Clopidogrel and 60-mg Prasugrel; Test type: Superiority or Other; p = 0.749, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 3]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.71, 95% CI 2-sided [-19.44 to 14.02]
Statistical Analysis 4: Comparison: Placebo and 60-mg Prasugrel vs 600-mg Clopidogrel and 30-mg Prasugrel; Test type: Superiority or Other; p = 0.890, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 3]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.15, 95% CI 2-sided [-15.24 to 17.53]
Statistical Analysis 5: Comparison: Placebo and 60-mg Prasugrel vs 600-mg Clopidogrel and 60-mg Prasugrel; Test type: Superiority or Other; p = 0.223, Mixed Model Repeated Measures Analysis — P-value is for 6 hours after prasugrel LD. P-values were not adjusted for multiplicity. P-values <0.05 were considered statistically significant; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -6.89, 95% CI 2-sided [-18.02 to 4.24]
Statistical Analysis 6: Comparison: Placebo and 60-mg Prasugrel vs 600-mg Clopidogrel and 30-mg Prasugrel; Test type: Superiority or Other; p = 0.808, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 5, analysis 5]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.33, 95% CI 2-sided [-9.44 to 12.10]
Statistical Analysis 7: Comparison: Placebo and 60-mg Prasugrel vs 600-mg Clopidogrel and 60-mg Prasugrel; Test type: Superiority or Other; p = 0.049, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 5]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -10.07, 95% CI 2-sided [-20.11 to -0.04]
Statistical Analysis 8: Comparison: Placebo and 60-mg Prasugrel vs 600-mg Clopidogrel and 30-mg Prasugrel; Test type: Superiority or Other; p = 0.842, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 5]; [statistical method as in outcome 1, analysis 1]; Median Difference (Final Values) = -0.99, 95% CI 2-sided [-10.85 to 8.86]
Statistical Analysis 9: Comparison: Placebo and 60-mg Prasugrel vs 600-mg Clopidogrel and 60-mg Prasugrel; Test type: Superiority or Other; p = 0.247, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 7]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -5.03, 95% CI 2-sided [-13.58 to 3.52]
Statistical Analysis 10: Comparison: Placebo and 60-mg Prasugrel vs 600-mg Clopidogrel and 30-mg Prasugrel; Test type: Superiority or Other; p = 0.942, Mixed Model Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 7]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.31, 95% CI 2-sided [-8.09 to 8.71]

6. Secondary Outcome: Percentage of Poor Responders
Description: Poor responders are those who had P2Y12 Reaction Units (PRU)≥ 240.
Time Frame: Baseline and 2 and 6 and 24 and 72 hours after loading dose
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Placebo and 60-mg Prasugrel | 600-mg Clopidogrel and 60-mg Prasugrel | 600-mg Clopidogrel and 30-mg Prasugrel
Number analyzed (Participants) | 52 | 47 | 50
percentage of participants
  Baseline | 68.1 | 66.7 | 51.2
  2 Hours after Prasugrel LD | 23.3 | 12.8 | 21.4
  6 Hours after Prasugrel LD | 11.6 | 5.3 | 4.4
  24 Hours after Prasugrel LD | 9.5 | 2.9 | 8.8
  72 Hours after Prasugrel LD | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: TEAE is a worsening or new occurrence of adverse event (AE) during treatment compared to baseline. A summary of serious adverse events (SAE) and other nonserious AE are located in the Reported Adverse Events section.
Time Frame: Baseline through 72 hours after prasugrel loading dose
Population: Participants who received any treatment.
Measure: Number; unit: participants
Arm/Group | Placebo and 60-mg Prasugrel | 600-mg Clopidogrel and 60-mg Prasugrel | 600-mg Clopidogrel and 30-mg Prasugrel
Number analyzed (Participants) | 109 | 79 | 88
participants
  Serious Adverse Events | 2 | 8 | 1
  Nonserious Adverse Events | 37 | 31 | 31

8. Secondary Outcome: P2Y12 Reaction Units (PRU) of Clopidogrel Treated Participants at Baseline by Cytochrome P450 2C19 (CYP2C19)-Predicted Functional Groups - CYP2C19 Extensive Metabolizers (EM) and Reduced Metabolizers (RM)
Description: CYP2C19 is a drug metabolizing enzyme. CYP2C19 Extensive metabolizers (EM) are individuals with two fully active / normal function CYP2C19 alleles (*1/*1, *1/*17). CYP2C19 Reduced metabolizers (RM) are individuals with at least one reduced-function CYP2C19 allele (*2/*2, *1/*2). Least Squares (LS) Mean values were controlled for CYP2C19 genetic group.
Time Frame: Baseline
Population: All randomized participants who were treated with Clopidogrel and had PRU measurement at Baseline and provided a DNA sample.
Measure: Least Squares Mean (Standard Error); unit: PRU
Groups:
- Clopidogrel at Baseline -CYP2C19 EM: 600-milligram (mg) clopidogrel loading dose (LD) administered once orally before percutaneous coronary intervention (PCI).
- Clopidogrel at Baseline - CYP2C19 RM: 600-mg clopidogrel LD administered once orally before PCI.
Arm/Group | Clopidogrel at Baseline -CYP2C19 EM | Clopidogrel at Baseline - CYP2C19 RM
Number analyzed (Participants) | 51 | 20
PRU | 243.549 (11.244) | 240.100 (17.955)
Statistical Analysis 1: Comparison: Clopidogrel at Baseline -CYP2C19 EM vs Clopidogrel at Baseline - CYP2C19 RM; A linear ANOVA model with PRU values at baseline for clopidogrel treated participants as response and CYP2C19 metabolizer status as covariate of main interest; Test type: Superiority or Other; p = 0.8711, ANOVA; Mean Difference (Final Values) = 3.449, 95% CI 2-sided [-38.81 to 45.71]

9. Secondary Outcome: P2Y12 Reaction Units (PRU) at 6 Hours Post-Prasugrel Loading Dose (LD) by Cytochrome P450 2C19 (CYP2C19)-Predicted Functional Groups - Extensive Metabolizers (EM) and Reduced Metabolizers (RM)
Description: as for outcome 8
Time Frame: 6 hours after prasugrel loading dose
Population: All randomized participants who received prasugrel LD and had PRU measurements 6 hours after prasugrel LD and provided a DNA sample.
Measure: Least Squares Mean (Standard Error); unit: PRU
Groups:
- Placebo and 60 mg Prasugrel-CYP2C19 EM: CYP2C19 extensive metabolizers treated with placebo loading dose (LD) administered once orally before percutaneous coronary intervention (PCI) and 60-milligram (mg) prasugrel LD administered once orally during PCI, followed by 10-mg prasugrel maintenance dose administered orally 24 hours after LD, then every 24 hours for 72 hours.
- Placebo and 60 mg Prasugrel -CYP2C19 RM: CYP2C19 reduced metabolizers treated with placebo LD administered once orally before PCI and 60-mg prasugrel LD administered once orally during PCI, followed by 10-mg prasugrel maintenance dose administered orally 24 hours after LD, then every 24 hours for 72 hours.
- 600 mg Clopidogrel and 60 mg Prasugrel - CYP2C19 EM: CYP2C19 extensive metabolizers treated with 600-mg clopidogrel LD administered once orally before PCI and 60-mg prasugrel LD administered once orally during PCI, followed by 10-mg prasugrel maintenance dose administered orally 24 hours after LD, then every 24 hours for 72 hours.
- 600 mg Clopidogrel and 60 mg Prasugrel - CYP2C19 RM: CYP2C19 reduced metabolizers treated with 600-mg clopidogrel LD administered once orally before PCI and 60-mg prasugrel LD administered once orally during PCI, followed by 10-mg prasugrel maintenance dose administered orally 24 hours after LD, then every 24 hours for 72 hours.
- 600 mg Clopidogrel and 30 mg Prasugrel - CYP2C19 EM: CYP2C19 extensive metabolizers treated with 600-mg clopidogrel LD administered once orally before PCI and 30-mg prasugrel LD administered once orally during PCI, followed by 10-mg prasugrel maintenance dose administered orally 24 hours after LD, then every 24 hours for 72 hours.
- 600 mg Clopidogrel and 30 mg Prasugrel - CYP2C19 RM: CYP2C19 reduced metabolizers treated with 600-mg clopidogrel LD administered once orally before PCI and 30-mg prasugrel LD administered once orally during PCI, followed by 10-mg prasugrel maintenance dose administered orally 24 hours after LD, then every 24 hours for 72 hours.
Arm/Group | Placebo and 60 mg Prasugrel-CYP2C19 EM | Placebo and 60 mg Prasugrel -CYP2C19 RM | 600 mg Clopidogrel and 60 mg Prasugrel - CYP2C19 EM | 600 mg Clopidogrel and 60 mg Prasugrel - CYP2C19 RM | 600 mg Clopidogrel and 30 mg Prasugrel - CYP2C19 EM | 600 mg Clopidogrel and 30 mg Prasugrel - CYP2C19 RM
Number analyzed (Participants) | 28 | 4 | 21 | 8 | 23 | 9
PRU | 39.036 (11.397) | 47.750 (30.153) | 20.190 (13.160) | 23.625 (21.321) | 36.478 (12.575) | 24.778 (20.102)
Statistical Analysis 1: Comparison: Placebo and 60 mg Prasugrel-CYP2C19 EM vs Placebo and 60 mg Prasugrel -CYP2C19 RM; A linear ANOVA model with PRU values of 6 hours post Prasugrel LD as response and treatment, CYP2C19 metabolizer status, interaction of treatment-by-CYP2C19 metabolizer status as fixed effects; Test type: Superiority or Other; p = 0.7875, ANOVA; Mean Difference (Final Values) = -8.714, 95% CI 2-sided [-72.78 to 55.36]
Statistical Analysis 2: Comparison: 600 mg Clopidogrel and 60 mg Prasugrel - CYP2C19 EM vs 600 mg Clopidogrel and 60 mg Prasugrel - CYP2C19 RM; A linear ANOVA model with PRU values of 6 hours Post-Prasugrel LD as response and treatment, CYP2C19 metabolizer status, interaction of treatment-by-CYP2C19 metabolizer status as fixed effects; Test type: Superiority or Other; p = 0.8913, ANOVA; Mean Difference (Final Values) = -3.435, 95% CI 2-sided [-53.23 to 46.37]
Statistical Analysis 3: Comparison: 600 mg Clopidogrel and 30 mg Prasugrel - CYP2C19 EM vs 600 mg Clopidogrel and 30 mg Prasugrel - CYP2C19 RM; [analysis description as in outcome 9, analysis 2]; Test type: Superiority or Other; p = 0.6229, ANOVA; Mean Difference (Final Values) = 11.700, 95% CI 2-sided [-35.43 to 58.83]

ADVERSE EVENTS:
Arm/Group | Placebo and 60-mg Prasugrel | 600-mg Clopidogrel and 60-mg Prasugrel | 600-mg Clopidogrel and 30-mg Prasugrel
Serious Adverse Events (participants affected / at risk) | 2/109 | 8/79 | 1/88
Other Adverse Events (participants affected / at risk) | 37/109 | 31/79 | 31/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo and 60-mg Prasugrel (N=109) | 600-mg Clopidogrel and 60-mg Prasugrel (N=79) | 600-mg Clopidogrel and 30-mg Prasugrel (N=88)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) — This event resulted in death after the participant had discontinued the study (participant decision).
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) — This event resulted in death.
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Femoral artery dissection (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo and 60-mg Prasugrel (N=109) | 600-mg Clopidogrel and 60-mg Prasugrel (N=79) | 600-mg Clopidogrel and 30-mg Prasugrel (N=88)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Angina pectoris (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 2 (2)
Chest pain (General disorders) | 1 (1) | 1 (1) | 2 (2)
Cardiac enzymes increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
High density lipoprotein decreased (Investigations) | 8 (8) | 7 (7) | 7 (7)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2)
Dyslipidaemia (Metabolism and nutrition disorders) | 5 (5) | 4 (4) | 2 (2)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 6 (6) | 3 (3) | 6 (6)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 3 (3) | 4 (4) | 4 (4)
Insomnia (Psychiatric disorders) | 0 (0) | 3 (3) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days